CLINICAL TRIAL: NCT06775015
Title: SERS-Based Serum Molecular Spectral Detection of Lung Cancer Microinvasion Versus Invasion Screening: A Multicenter, Open-Label, Double-Blind, Independent Data Analysis Clinical Trial
Brief Title: SERS-Based Serum Molecular Spectral Detection of Invasive Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-043
Record Dates: First submitted 2025-01-05; First posted 2025-01-14 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer Patients
Keywords: SERS，Raman，Early screening for lung cancer，Pulmonary nodule，diagnostic model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who underwent chest CT scans and were found to have lung nodules: Chest CT confirmed the presence of pulmonary nodules in the patient and ultimately underwent surgical intervention. The pulmonary nodules had the final pathological results.
  Interventions: Diagnostic Test: Serum Raman spectroscopy intelligent diagnostic system

INTERVENTIONS:
Diagnostic Test: Serum Raman spectroscopy intelligent diagnostic system — Serum Raman spectroscopy intelligent diagnostic system Description: 1. Screening interested participants should sign the appropriate informed consent (ICF) prior to completion any study procedures. 2. The investigator will review symptoms, risk factors, and other non-invasive inclusion and exclusion criteria. 3. The following is the general sequence of events during the 3 months evaluation period: 4. Completion of baseline procedures Participants were assessed for 3 months and completed all safety monitoring.

SUMMARY:
Surgery is the main treatment for early lung cancer. It is worth noting that there are significant differences in postoperative prognosis and surgical methods between microinvasive cancer and early-stage invasive cancer. Micro invasive lung cancer can achieve 100% long-term survival through surgical resection, without the need for postoperative adjuvant radiotherapy. There is no need to remove lung lobes during surgery, only segmental or wedge resection is required, and systematic lymph node dissection is not recommended. Therefore, accurate prediction of preoperative and intraoperative microinvasive cancer and invasive cancer in pulmonary nodules is crucial for patients to choose surgical methods, which can significantly affect postoperative lung function retention and overall survival.

Raman spectroscopy (RS), as a non-invasive and highly specific molecular detection technique, can be obtained at the molecular level to sensitively detect changes in biomolecules composed of proteins, nucleic acids, lipids, and sugars related to tumor metabolism in biological samples. The surface enhanced Raman spectroscopy (SERS) developed based on this technology is one of the feasible methods for high-sensitivity biomolecule analysis.

We collected serum Raman spectroscopy data from a cohort of 138 early lung cancer patients in our preliminary research. Based on a machine learning model, we constructed an early lung microinvasive cancer and invasive cancer Raman intelligent diagnosis system, which achieved an accuracy rate of 89.4%. To obtain the highest level of clinical evidence and truly achieve clinical translation, this prospective, multicenter clinical study aims to validate the use of this intelligent diagnostic system for early diagnosis of lung cancer and the discrimination between microinvasive cancer and invasive cancer.

DETAILED DESCRIPTION:
1. Screening interested participants should sign the appropriate informed consent (ICF) prior to completion any study procedures.
2. The investigator will review symptoms, risk factors, and other non-invasive inclusion and exclusion criteria.
3. Completion of baseline procedures, participants were assessed for 30 days and completed all safety monitoring.
4. After completing the baseline assessment and confirming enrollment, participants will be given 2ml of fasting venous blood.

ELIGIBILITY:
Inclusion Criteria:

1. Participants confirmed by chest CT to have pulmonary nodules
2. The diagnosis of participants with malignant pulmonary nodules must meet the TNM diagnostic criteria (Ninth Edition);
3. Participants are willing to participate in this study and follow the research plan;
4. Participants or legally authorized representatives can give written informed consent approved by the Ethics Review Committee that manages the website;

Exclusion Criteria:

1. Participants with concomitant other malignant tumors;
2. Participants with missing baseline clinical data;
3. Participants with severe underlying lung diseases (such as bronchiectasis, bronchial asthma or COPD, etc.), or those with a history of occupational or environmental exposure to dust, mines or asbestos;
4. Participants who do not cooperate or refuse to participate in clinical trials at a later stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chest CT reveals the presence of pulmonary nodules in the patient and plans to undergo surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-04-04 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | through study completion, an average of 1 year
  Determine whether there is hematogenous metastasis in enrolled lung cancer patients through RAMAN intelligent diagnostic system
Time to RAMAN diagnosis | up to 30 days
  The time to perform RAMAN testing and obtain diagnostic results after obtaining serum

SECONDARY OUTCOMES:
Safety assessment Results | up to 30 days
  AEs and SAEs through Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- The 900th Hospital of the Joint Logistic Support Force, PLA, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes